CLINICAL TRIAL: NCT03419845
Title: A Pilot Investigation Into Frequent Fallers' Experiences of an Adapted Walking Frame, Designed to Reduce the Walking Aid's Associated Falls Risk
Brief Title: Frequent Fallers' Experiences of an Adapted Walking Frame, Designed to Reduce the Walking Aid's Associated Falls Risk
Acronym: Walker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham Community Healthcare NHS (Other Government)
Collaborators: Birmingham City University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 216488
Record Dates: First submitted 2017-02-20; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Falls Injury

STUDY DESIGN:
Intervention Model Description: Single arm, open trial to qualitatively explore the user's experience of the Step Right Buddy after a one week pilot trial and to assess the introduction of new risks to the patient as a result of the adaptation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Step Right Buddy arm (Experimental): To use modified walking frame using the Step Right Buddy
  Interventions: Device: Step Right Buddy

INTERVENTIONS:
Device: Step Right Buddy — The Step Right Buddy, which is under investigation in this clinical study, is an elasticated band that attached by Velcro to the back legs of a standard walking frame. The purpose of the Step Right Buddy is to provide sensory feedback to standard walking frame users of how far to step in to the frame and to encourage them to move the frame forward.

SUMMARY:
For some patients with mobility issues, a walking frame (commonly known as a zimmer frame - trademark of Zimmer Holdings), is provided to keep them on their feet and help them remain more independent in their home and when out and about. When patients are given the walking frame, they are given information on how to use it safely to protect them from hurting themselves. For a small group of patients, using the walking frame is difficult, and they will have a fall because they are unable to use the frame safely. For these patients, a fear of falling can then develop and they can then have more falls. It is thought that these falls with the walking frame happen because the patient steps too far into the frame, making them unstable. We have made an attachment for a standard walking frame, which we are calling the Step Right Buddy, that we think will help improve the stability of patients who step too far into the frame. We have attached a detachable elasticated band across the back legs of the frame to make patients aware that they have stepped far enough into the frame, to stop them stepping any further. In order to develop this further, we need to understand how people feel using this adapted frame and whether there are any new risks to the user.

The investigators propose to ask patients who are considered to be at risk of falling because of the way they use their walking frame if they would like to use the adapted walking frame in their home, instead of their standard frame, for a week. At the end of this week, investigators will spend up to an hour with this patient, talking with them about their experience of the adapted walking frame, in order to understand things such as how they felt using the frame, were they more or less fearful of using it than their usual frame, did they think they were going to fall over more or less often, do they think they fall more or less often. In addition to this, patients will keep a written record of when they thought they nearly fell, or when they had an injury whilst using the adapted walking frame. This information will be used to explore whether or not the adaption to the frame introduces new risks to patients.

DETAILED DESCRIPTION:
Title: A pilot investigation into frequent fallers' experiences of an adapted walking frame, designed to reduce the walking aid's associated falls risk.

Short title: The Walker Study

Chief Investigator: Dr Sarahjane Jones

Objectives:

To qualitatively explore the user's experience of the Step Right Buddy after a one week pilot trial and to assess the introduction of new risks to the patient as a result of the adaptation.

Trial configuration:

Qualitatively assessed clinical trial of a novel product.

Setting: Community care - patient homes.

Sample size: 20

Description of intervention: Application of the Step Right Buddy to the standard walking frame for patients to use as normal at home for one week.

Study duration:

Project length: March 2017 - July 2017

Length of participation - 1 week from consent

Randomisation and blinding: Single arm, open trial

Outcome measures: Participants' experiences of using the Step Right Buddy and adverse event data.

Analysis techniques: Framework analysis of textual data regarding the participants experiences and, where appropriate, root cause analysis of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Purposively sampled as those identified as 'fallers' as a result of their use of the walking frame or at risk of falling currently on the case load of the rehabilitation team within Birmingham Community Healthcare NHS Trust
* Routinely use walking frame to manoeuvre around the house and/or outside
* 18 years old or greater (no upper age limit)
* Have no visual impairments
* Must have mental capacity to consent for themselves
* Must speak, read and comprehend English to participate in the interview

Exclusion Criteria:

* This are not perceived to be at risk of falling as a result of their use of the walking frame
* Are younger than 18 years of age
* Are visually impaired
* Do not have mental capacity to consent for themselves
* Cannot comprehend written and spoken English sufficiently to give informed consent
* Are unable to follow the safety instructions for using the Step Right Buddy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
User experience | 1 week
  User experience will be assessed by asking the patient to trial the attachment for one week, completing a risk form during this week and providing verbal feedback at the end of this week.

SECONDARY OUTCOMES:
Adverse events | 1 week
  To assess the introduction of new risks to the patient as a result of the adaptation

CONTACTS AND LOCATIONS:
Overall Officials: Sarahjane Jones, PhD, Principal Investigator — Honorary contract - Birmingham Commnity Healthcare NHS Foundation Trust (substantive post with Birmingham City University)
Locations (1):
- Clive Thursfield, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
NA we are not making IPD available to other researchers.